CLINICAL TRIAL: NCT06430866
Title: A Randomized, Double-blind Study to Compare the Pharmacokinetics Between ABP 234 and Keytruda® (Pembrolizumab) in Participants With Early-stage Non-squamous Non-small Cell Lung Cancer as Adjuvant Treatment Following Resection and Platinum-based Chemotherapy
Brief Title: Pharmacokinetic Similarity Between ABP 234 and Keytruda® (Pembrolizumab)
Acronym: Eucalyptus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230127
Record Dates: First submitted 2024-03-15; First posted 2024-05-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Early-stage Non-squamous Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Keytruda; Pembrolizumab; ABP 234
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABP 234 (Experimental): Participants will receive ABP 234 every 3 weeks (Q3W) for up to 12 months.
  Interventions: Drug: ABP 234
- Pembrolizumab (Active Comparator): Participants will receive pembrolizumab Q3W for up to 12 months.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: ABP 234 — Administered by intravenous (IV) injection.
  Arms: ABP 234
Drug: Pembrolizumab — Administered by IV injection.
  Arms: Pembrolizumab

SUMMARY:
The primary objective of this study is to demonstrate pharmacokinetic (PK) similarity ABP 234 with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age.
* Pathological diagnosis of non-squamous NSCLC.
* Stage IB (T2 ≥ 4 cm), II, or IIIA NSCLC after complete surgical resection and received platinum-based chemotherapy.
* For programmed death-ligand 1 (PD-L1) testing, tumor tissue from the resected site of disease must be sent, received, and analyzed for biomarkers.
* Treated with platinum-based chemotherapy:

  1. Chemotherapy must have begun within 12 weeks after the resection surgery.
  2. The last chemotherapy dose must have been completed at least 3 weeks and no more than 12 weeks before the participant is randomized.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
* Epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), and ROS-1 negative.
* Have adequate organ function as indicated by laboratory values.
* Absence of severe comorbidities that in the opinion of the investigator might hamper participation in the study and/or treatment administration.
* Participants must sign approved informed consent form (ICF).

Exclusion Criteria:

* Evidence of disease.
* Prior treatment with anti-programmed cell death protein 1 and anti-PD-L1/2 modulating agents in adjuvant setting.
* History or presence of immune-mediated disorders.
* Participants with type 1 diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders not requiring systemic treatment are permitted to enroll.
* Participant has positive screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C (HCV).
* History of congenital immunodeficiency diseases, prior allogeneic stem cell transplantation, or organ transplantation.
* History of any other malignancy other than NSCLC within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, papillary thyroid cancer treated with surgery, etc.
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis virus, current alcohol abuse or cirrhosis.
* Surgery or chemotherapy-related toxicity not resolved to grade 1 with the exception of grade ≤ 2 alopecia, fatigue, neuropathy, and lack of appetite/nausea.
* Woman of childbearing potential who is pregnant or is breast feeding.
* Woman of childbearing potential who is not consenting to use highly effective methods of birth control.
* Man with a partner of childbearing potential who does not consent to use highly effective methods of birth control.
* Participant has known hypersensitivity to monoclonal antibodies or to any of the excipients of the investigational product (IP).
* Active cardiac disease or history of cardiac dysfunction, that in the judgment of the investigator would place the participant at additional risk when participating in the study.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current neumonitis/interstitial lung disease.
* Live vaccine therapy within 4 weeks prior to IP administration.
* Participation in another investigational drug study within 30 days prior to IP administration.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve (AUC) From Time 0 to 21 Days (AUC21d) Following the First Dose | 21 days
AUC at Steady State Between Week 16 and Week 19 (AUCtau_ss) | Weeks 16-19

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) Following the First Dose (Cmax_dose1) | Up to 65 weeks
Time to Maximum Serum Concentration (Tmax) Following the First Dose (Tmax_dose1) | Up to 65 weeks
Cmax at Steady State (Cmax_ss) | Weeks 16-19
Tmax at Steady State (Tmax_ss) | Weeks 16-19
Trough Serum Concentrations (Ctrough) at Pre-dose of Week 4 (Ctrough_w4) | Week 4 pre-dose
Ctrough at Stead State (Ctrough_ss) | Weeks 16 and 19 pre-dose
Number of Participants with Treatment-emergent Adverse Events | Up to 16 months
Number of Participants with Treatment-emergent Serious Adverse Events | Up to 16 months
Number of Participants with Treatment-emergent Adverse Events of Interest (EOIs) | Up to 16 months
Number of Participants with Andit-drug Antibodies | Baseline and weeks 4, 7, 16, 19, 22, 28, 40, 52, and 65
Disease-free Survival | Up to 65 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (128):
- Argentina (3):
  - Fundacion ARS Medica, San Salvador de Jujuy, Jujuy Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Ionc Instituto Oncologico De Cordoba, Córdoba
- University Multiprofile Hospital for Active Treatment Sofiamed, Sofia, Bulgaria
- Chile (8):
  - CDIEM - Centro de Investigacion y Especialidades Medicas, Providencia, Region Metropolotana
  - Centro de Investigaciones Clinicas Vina del Mar Ltda., ViÃ±a Del Mar, Región de Valparaíso
  - Centro de Investigacin de Enfermedades Respiratorias e Inmunologicas Limitada CIERI, Viña del Mar, Región de Valparaíso
  - Instituto Oncologico Fundacion Arturo Lopez Perez (FALP), Providencia, Santiago Metropolitan
  - Centro de Oncologa de Precisin, Region Metropolitana, Santiago Metropolitan
  - Clinica Santa Maria, Santiago, Santiago Metropolitan
  - K2 Oncology, Santiago
  - Icegclinic Research and Care, Santiago
- France (7):
  - Clinique Belharra Ramsay Sante, Bayonne
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint - Andre, Bordeaux
  - Centre Francois Baclesse, Caen
  - Hopital Europeen Marseille, Marseille
  - Hopital Bichat, APHP, Paris
  - Centre Hospitalier Intercommunal Toulon La Seyne Sur Mer (C.H.I.T.S) - Hopital Sainte Musse, Toulon
  - Hopital Robert Schuman, Vantoux
- Georgia (2):
  - LLC Todua Clinic, Tbilisi
  - New Hospitals, Tbilisi
- Germany (2):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Kliniken Essen Mitte, Evang. Huyssens-Stiftung, Internistische Onkologie und Hmatologie mit integire, Essen
- Italy (12):
  - Azienda Ospedaliero - Universitaria di Ferrara, Cona
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Versilia, Lucca
  - Azienda USL 2 Lucca, Lucca
  - AOU Cagliari-Policlinico Universitario Duilio Casula di Monserrato-UOC Oncologia Medica, Monserrato
  - ASL Napoli 1 Centro-Ospedale del Mare, Napoli
  - Casa Di Cura Polispecialistica Dott Pederzoli, Peschiera del Garda
  - AUSL Della Romagna - Ospedale S.Maria delle Croci, Ravenna
  - IRCCS Istituto clinico humanitas - Humanitas Mirasole spa, Rozzano
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - ASST Sette Laghi, Varese
- Malaysia (3):
  - Raja Perempuan Zainab II Hospital, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching, Sarawak
- Mexico (7):
  - Preparaciones Oncolgicas S.C., LeÃ³n, Guanajuato
  - Investigacion Biomedica para el Desarrollo de Nuevos Farmacos SA de CV, Zapopan, Jalisco
  - Centro Medico Dalinde, Cuauhtémoc, Mexico City
  - Accelerium Clinical Research, Monterrey, Nuevo León
  - Onco Pall Advance Care Oncology Center Sa de CV, Monterrey, Nuevo León
  - iCan Oncology Center S.A. de C.V., Monterrey, Nuevo León
  - Clinica Integral Internacional de Oncolgia S de RL de CV, Puebla City
- Philippines (6):
  - Cebu Doctors University Hospital, Cebu City, Cebu
  - Davao Doctors Hospital, Davao City, Davao Del Sur
  - Makati Medical Center, Makati City, National Capital Region
  - Veterans Memorial Medical Center, Quezon City, National Capital Region
  - Riverside Medical Center Inc, Bacolod City, Negros Occidental
  - Philippine General Hospital, Manila
- Poland (6):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Warminsko Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o, Krakow
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - Gyncentrum Szpital, Sosnowiec
- Romania (5):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - Oncocenter Oncologie Clinica S.R.L, Timișoara, Timiș County
  - Oncomed, Timișoara, Timiș County
  - S.C. Medisprof S.R.L, Cluj-Napoca
  - Centrul de Oncologie Euroclinic srl, Jud. Iasi
- Serbia (2):
  - Clincial Centre of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
- South Korea (11):
  - The Catholic University Of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Pusan National University Hospital (PNUH), Busan
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center (AMC), Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (25):
  - Centro Oncologico de Galicia, A Coruna Galicia
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Universitario de Elche, Alicante
  - Institut Catala d'Oncologia Badalona, Hospital Germans Trias I Pujol, Badalona
  - UOMI Cancer Center-Clinica Tres Torres, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Quiron Dexeus Barcelona, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Hospital Universitario San Francisco de Asis, Madrid
  - Clinica MD Anderson International, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Unifersitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital De Mataro, Mataró
  - Hospital Quironsalud Malaga, MÃ¡laga
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Complejo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario De Valme, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulev, Valencia
  - Hospital Clinico Univ Valladolid, Valladolid
- Taiwan (6):
  - National Taiwan University Hospital (NTUH), Taipei, Zhongzheng Dist
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung County
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (7):
  - Mahidol University - Siriraj Hospital - Siriraj Clinical Research Center (SICRC), Bangkoknoi, Bangkok
  - King Chulalongkorn Memorial Hospital, Chulalongkom University, Pathumwan, Bangkok
  - Lampang Cancer Hospital, Muang, Changwat Lampang
  - Naresuan University Hospital, Muang, Changwat Phitsanulok
  - Prince Of Songkla Hospital, Prince Of Songkhla University, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Muang, Chiang Mai
  - Faculty of Medicine Vajira Hospital, Navamindradhiraj University, Bangkok
- Turkey (Türkiye) (15):
  - Gazi University Faculty of Medicine, Yenimahalle, Ankara
  - Trakya University Faculty of Medicine, İskender, Edirne
  - Medical Park Seyhan Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Baskent University Ankara Hospital, Ankara
  - Uludag University Faculty of Medicine, Bursa
  - Medical Point Gaziantep Hospital, Gaziantep
  - Bezmialem Foundation University Medical Faculty, Istanbul
  - Sakarya University - Faculty of Medicine, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com